CLINICAL TRIAL: NCT00167141
Title: Hormonal Male Contraception in Men With Normal and Subnormal Semen Parameters
Brief Title: Contraception in Normal and Subnormal Men
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Prof. Dr. Eberhard Nieschlag, University Hospital Muenster
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRM 2003/21; IRM 2003/21
Record Dates: First submitted 2005-09-06; First posted 2005-09-14 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2007-03

CONDITIONS: Healthy
Keywords: male fertility; semen parameters

ARMS (1):
- testosterone injections (Experimental): injections of testosterone to normal men (arm 1) and two men with subnormal semen parameters (arm 2)
  Interventions: Drug: injection of hormonal male contraceptive

INTERVENTIONS:
Drug: injection of hormonal male contraceptive — testosterone injections 4 times

SUMMARY:
Volunteers with normal and subnormal semen parameters receive a hormonal male contraceptive in order to investigate whether there are differences between normal and subnormal men in terms of suppressibility, rate of azoospermia and reversibility of suppression of spermatogenesis.

DETAILED DESCRIPTION:
Volunteers with normal and subnormal semen parameters receive a hormonal male contraceptive in order to investigate whether there are differences between normal and subnormal men in terms of suppressibility, rate of azoospermia and reversibility of suppression of spermatogenesis. Twenty-five men will be recruited for each group. They will be exposed to hormonal male contraception for six months.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with normal and subnormal semen parameters

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
semen parameters | 2005 - 2008

SECONDARY OUTCOMES:
hormones | 2005 2008

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Nieschlag, Prof. Dr., Principal Investigator — Institute of Reproductive Medicine
Locations (1):
- Prof. Dr. Eberhard Nieschlag, Münster, Germany